CLINICAL TRIAL: NCT02958189
Title: Tweet4Wellness: An Online Virtual Support Group for Promoting Increased Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Judith Prochaska, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32127
Record Dates: First submitted 2016-02-22; First posted 2016-11-08 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Physical Activity; Social Media
Keywords: Twitter; social support; internet intervention; sedentary lifestyle; walking; behavior change
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Tweet4Wellness+Self-monitoring (Experimental): This group will receive the Tweet4Wellness intervention: daily theory-based peer-to-peer discussion prompt within the private Twitter-based support group for the entire 6 months of the study. They will also receive the Fitbit triaxial pedometer that will track their daily steps (self-monitoring component).
  Interventions: Behavioral: Tweet4Wellness; Behavioral: Self-monitoring
- Group 2: Self-monitoring (Active Comparator): This group will receive the Fitbit triaxial pedometer that will track their daily steps (self-monitoring component) for the first 3 months. For the second three months of the study, they will receive the Tweet4Wellness intervention in addition to their Fitbit self-monitoring.
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Tweet4Wellness — A daily, behavior change theory-based intervention message is sent to a private, 25-person online Twitter-support group to prompt peer-to-peer discussion. Participants receive individual text messages to encourage group participation (e.g. 'thank you for participating' or 'please participate tomorrow'). Participants also receive weekly individual messages giving them daily step goals for the week based on their previous week's daily step average, recorded from Fitbit.
  Arms: Group 1: Tweet4Wellness+Self-monitoring
Behavioral: Self-monitoring — A Fitbit is provided to the group which tracks participants' daily steps.

SUMMARY:
The purpose of this study is to determine whether a Twitter-based intervention with a private, online support group can significantly increase number of walking steps compared to self-monitoring of physical activity alone or a control group in sedentary women at a women's heart clinic.

DETAILED DESCRIPTION:
Sedentary behavior is a risk factor for heart disease, independent of meeting physical activity guidelines. Tweet4Wellness is an innovative light physical activity, specifically walking, intervention which randomly assigns participants to a 25-person private, online support group that will receive daily, theory-based messages as peer-to-peer discussion prompts. Many text-based interventions do not base the intervention text messages in behavior change theory, but this study will base the daily messages in the behavior change theories such as implementation intentions, social support, mindfulness, and social learning theory.

The trial will be conducted over a 6-month periods. For the first 3 months, there will be 2 groups: Group 1 will receive the Twitter intervention and a "Fitbit" triaxial pedometer to track their steps throughout the day; Group 2 will receive the Fitbit pedometer only.

For the second 3 months: Group 1 an Group 2 will track their physical activity with Fitbit only.

ELIGIBILITY:
Inclusion Criteria:

* Are a woman
* Are over 18 years of age
* Are English speaking
* Have or are willing to purchase a mobile phone with a camera
* Have or are willing to purchase an unlimited text plan
* Are willing to participate in daily tweets or texts for up to 3 months
* Have an active email account
* Have internet access on your mobile phone
* Use or are familiar with Facebook, Twitter, or other social media
* Text at least weekly

Exclusion Criteria:

* Have certain symptoms or conditions that would not be conducive to increasing your physical activity as determined by your physician
* Are planning on becoming pregnant in the next 8 months
* If our screening survey indicates that you are already adequately physically active
* Do not provide all required personal contact information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in steps (physical activity) | Baseline to 3 months and 6 months
  Steps measured by triaxial accelerometer

SECONDARY OUTCOMES:
Support Group Engagement during the intervention | 3 months
  Measured by # of Tweets per day sent to the group
average length of prolonged sedentary periods per day | baseline to 3 months and 6 months
  average length of uninterrupted sedentary periods per day over a seven day period

CONTACTS AND LOCATIONS:
Overall Officials: Judith Prochaska, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Oppezzo M, Tremmel J, Desai M, Baiocchi M, Ramo D, Cullen M, Prochaska JJ. Twitter-Based Social Support Added to Fitbit Self-Monitoring for Decreasing Sedentary Behavior: Protocol for a Randomized Controlled Pilot Trial With Female Patients From a Women's Heart Clinic. JMIR Res Protoc. 2020 Dec 4;9(12):e20926. doi: 10.2196/20926. PMID 33275104